CLINICAL TRIAL: NCT00039026
Title: A Phase 3, Randomized, Triple-Blind, Parallel-Group, Long-Term, Placebo-Controlled, Multicenter Study to Examine the Effect on Glucose Control (HbA1c) of AC2993 Given Two Times a Day in Subjects With Type 2 Diabetes Mellitus Treated With a Sulfonylurea Alone
Brief Title: Evaluation of the Effect on Glucose Control of AC2993 in Patients With Type 2 Diabetes Mellitus Treated With a Sulfonylurea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2993-113
Record Dates: First submitted 2002-06-06; First posted 2002-06-10 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Type 2 Diabetes Mellitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AC2993 5 mcg (0.02 mL) (Experimental): Placebo, then AC2993 5 mcg, then AC2993 5 mcg
  Interventions: Drug: AC2993
- AC2993 10mcg (0.04 mL) (Experimental): Placebo, then AC2993 5 mcg, then AC2993 10 mcg
  Interventions: Drug: AC2993
- Placebo 0.02 mL (Placebo Comparator): Placebo 0.02 mL, then Placebo 0.02 mL, then Placebo 0.02 mL
  Interventions: Drug: Placebo
- Placebo 0.04 mL (Placebo Comparator): Placebo 0.02 mL / Placebo 0.02 mL / Placebo 0.04 mL
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AC2993 — Placebo Lead In (0.02 mL) for 4 weeks / AC2993 5mcg (0.02 mL) for 4 weeks / AC2993 5mcg (0.02 mL) for 26 weeks - All are subcutaneously injected twice daily
  Other Names: synthetic exendin-4
  Arms: AC2993 5 mcg (0.02 mL)
Drug: AC2993 — Placebo Lead In (0.02 mL) for 4 weeks / AC2993 5mcg (0.02 mL) for 4 weeks / AC2993 5mcg (0.02 mL) for 26 weeks - All are subcutaneously injected twice daily
  Other Names: synthetic exendin-4
  Arms: AC2993 10mcg (0.04 mL)
Drug: Placebo — Placebo Lead In (0.02 mL) for 4 weeks / Placebo (0.02 mL) for 4 weeks / Placebo (0.02 mL) for 26 weeks - All are subcutaneously injected twice daily
  Arms: Placebo 0.02 mL
Drug: Placebo — Placebo Lead In (0.02 mL) for 4 weeks / Placebo mcg (0.02 mL) for 4 weeks / Placebo (0.04 mL) for 26 weeks - All are subcutaneously injected twice daily
  Arms: Placebo 0.04 mL

SUMMARY:
This is a multicenter, randomized, blinded, placebo-controlled study to assess the effects on glucose control of AC2993 as compared to placebo in patients with type 2 diabetes. Patients will be randomized into one of two AC2993 treatment arms or to placebo treatment and will continue with their required existing diabetes medication (sulfonylurea) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 diabetes mellitus
* Treated with a sulfonylurea at defined doses for at least 3 months prior to screening
* BMI= 27-45 kg/m2
* HbA1c value between 7.5% and 11%

Exclusion Criteria:

* Treated with oral anti-diabetic medications other than a sulfonylurea within 3 months of screening
* Patients treated previously with AC2993
* Patients presently treated with insulin

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2002-02; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from Baseline to Week 30 | Baseline (Day 1) to Week 30
  Change in HbA1c from Baseline (Day 1) to study termination (Week 30)

SECONDARY OUTCOMES:
Change in HbA1c from baseline (Day 1) to each of the intermediate visits | Baseline (Day 1), Week 2, Week 4, Week 6, Week 12, Week 18, Week 24
  Change in HbA1c from baseline, measured from Visit 3 (Day 1) to each of the intermediate visits (Baseline (Day 1), Week 2, Week 4, Week 6, Week 12, Week 18, and Week 24
The number of subjects achieving HbA1c target values of < 7% and < 8% by Week 30 | Baseline (Day 1) and Week 30
  The number of subjects achieving HbA1c target values of < 7% and < 8% by study termination (Week 30)
The number of subjects achieving HbA1c reductions of > 0.5% and > 1.0% by Week 30 | Baseline (Day 1), and Week 30
  The number of subjects achieving HbA1c reductions of > 0.5% and > 1.0% by study termination (Week 30)
The time to achieve HbA1c reductions of 0.5% or more and >1.0% or more | Baseline (Day 1), Week 2, Week 4, Week 6, Week 12, Week 18, Week 24, Week 30
  The time it takes subjects to achieve HbA1c reductions of 0.5% or more and >1.0% or more
The time to achieve specific HbA1c target values of < 7% and < 8% | Baseline (Day 1), Week 2, Week 4, Week 6, Week 12, Week 18, Week 24, Week 30
  The time it takes subjects to achieve HbA1c target values of < 7% and < 8%
Change in body weight from Baseline to each intermediate visit and Week 30 | Baseline (Day 1), Week 2, Week 4, Week 6, Week 12, Week 18, Week 24, Week 30
  Change in body weight (kg) from Baseline to each intermediate visit and Week 30

CONTACTS AND LOCATIONS:
Locations (126):
- United States (126):
  - Pinnacle Research Group, Anniston, Alabama
  - Parkway Medical Center, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Eclectic Family Care, Eclectic, Alabama
  - Winston Physician Services, Haleyville, Alabama
  - Simon Williamson Clinic, Hueytown, Alabama
  - Extended Arm Physicians/ Southern Drug, Montgomery, Alabama
  - Southern Drug Research Network, Tallassee, Alabama
  - Clinic of Physicians and Surgeons, Ltd., Mesa, Arizona
  - ANA Ventures, LLC, Mesa, Arizona
  - Lovelace Scientific Resources-Phoenix, Phoenix, Arizona
  - Physicians at the Peak, Phoenix, Arizona
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - CAVHS, Little Rock, Arkansas
  - Physicians Group Research Clinic, LLC, Little Rock, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - Mitchell Research Group, Inc., Bakersfield, California
  - William Zigrang, M.D., Burlingame, California
  - International Clinical Research Network, Chula Vista, California
  - Arrowhead Regional Medical Center, Colton, California
  - East Bay Clinical Trial Center, Concord, California
  - Valley Research, Fresno, California
  - Tushar Modi, M.D., Modesto, California
  - Elke Jost-Vu, M.D., Rancho Mirage, California
  - Comprehensive Diabetes-Endocrine Medical Associates, Redwood City, California
  - nTouch, San Diego, California
  - Radiant Research-San Diego, San Diego, California
  - Veterans Medical Research Foundation, San Diego, California
  - Diabetes Research Institute of Mills Peninsula, San Mateo, California
  - Advanced Clinical Research Institute, Santa Ana, California
  - West Coast Clinical Trials, Signal Hill, California
  - Protocare Trials at Sharp Mission Park, Vista, California
  - Diablo Clinical Research, Walnut Creek, California
  - George Washington University, Washington D.C., District of Columbia
  - Internal Medicine Associates, Fort Myers, Florida
  - Clin Sci International, Gainesville, Florida
  - University of FL, Gainesville, Florida
  - Jupiter Research Institute, Jupiter, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - Tampa Medical Group, Tampa, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Radiant Research, West Palm Beach, Florida
  - Clinical Research Atlanta, Atlanta, Georgia
  - nTouch Research Corporation, Decatur, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - St. Luke's Family Health, Meridian, Idaho
  - University Primary Care Center at Belvidere, Belvidere, Illinois
  - Northwestern Memorial Physicians Group, Chicago, Illinois
  - Illinois Center for Clinical Trials, Chicago, Illinois
  - Medical Group of Fort Wayne, Fort Wayne, Indiana
  - American Health Network, Indianapolis, Indiana
  - nTouch Research-South Bend, South Bend, Indiana
  - Kentucky Diabetes Center, Lexington, Kentucky
  - University of Kentucky Metabolic Research Group, Lexington, Kentucky
  - MedResearch, Inc., Louisville, Kentucky
  - Drug Research Services, Metairie, Louisiana
  - New Orleans Institute of Clinical Investigation, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - St. Agnes Health Care, Baltimore, Maryland
  - Doctors Research Associates of Maryland, Lanham, Maryland
  - Grunberger Diabetes Medical Center, Bloomfield Hills, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Grand Rapids Associated Interns, Grand Rapids, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Diabetes and Endocrinology Specialists, Chesterfield, Missouri
  - Midwest Pharmaceutical Research, City of Saint Peters, Missouri
  - Mid Missouri Research Specialists, Inc., Rolla, Missouri
  - Radiant Research-St. Louis, St Louis, Missouri
  - Mercury Street Medical, Butte, Montana
  - Lovelace Scientific Resources-Las Vegas, Las Vegas, Nevada
  - HIS Clinical Research, Jersey City, New Jersey
  - Radiant Research-Moorestown, Moorestown, New Jersey
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Medical Network Services, P.C., Brooklyn, New York
  - St. Lukes Roosevelt Hospital, New York, New York
  - Naomi Berrie Diabetes Center at Columbia University, New York, New York
  - Heights Medical Care, New York, New York
  - DOCS at Beth Israel Medical Center, Yonkers, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Charlotte Clinical Research, Charlotte, North Carolina
  - UNC Diabetes Care Center, Durham, North Carolina
  - Unifour Medical Research, Hickory, North Carolina
  - New Hanover Medical Research Associates, Wilmington, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Rapid Medical Research, Cleveland, Ohio
  - Ohio State University-Division of Endocrinology, Columbus, Ohio
  - Radiant Research-Columbus, Columbus, Ohio
  - University Mednet, Mentor, Ohio
  - Comprehensive Research Services, Inc., Mogadore, Ohio
  - COR Clinical Research, Oklahoma City, Oklahoma
  - nTouch Research Corporation-Oklahoma City, Oklahoma City, Oklahoma
  - Utica Park Clinic, Tulsa, Oklahoma
  - Medford Medical Clinic, Medford, Oregon
  - Legacy Clinical Research, Portland, Oregon
  - Radiant Research, Portland, Oregon
  - Physicians for Clinical Research, Camp Hill, Pennsylvania
  - Thomas Jefferson University Diabetes Research Center, Philadelphia, Pennsylvania
  - Philadelphia Health Associates, Philadelphia, Pennsylvania
  - Tipton Medical and Diagnostic Center, Tipton, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Radiant Research-Charleston, Charleston, South Carolina
  - CNS Clinical Trials, Chester, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Integrity Clinical Research, Jackson, Tennessee
  - Harmony Clinical Research, Johnson City, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Endocrine Consultants of ET, Knoxville, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - Texas Tech University Health Sciences-Internal Medicine, El Paso, Texas
  - Internal Medicine Associates, El Paso, Texas
  - North Texas Clinical Research, Irving, Texas
  - Dr. Humberto Bruschetta, Kingsville, Texas
  - South Texas Applied Research, McAllen, Texas
  - University of Texas Health Sciences Center-Texas Diabetes Institute, San Antonio, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
  - SAM Clinical Research Center, San Antonio, Texas
  - Salt Lake Research, Salt Lake City, Utah
  - Clinical Research Center-Eastern Virginia Medical School, Norfolk, Virginia
  - West Olympia Internal Medicine, Olympia, Washington
  - Rainier Clinical Research Center, Renton, Washington
  - Northside Internal Medicine, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Julia M. Hutchinson, M.D., Spokane, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - Hyperion Clinical Research, Charleston, West Virginia
  - CAMC Clinical Trials Center, Charleston, West Virginia

REFERENCES:
- [Result] Buse JB, Henry RR, Han J, Kim DD, Fineman MS, Baron AD; Exenatide-113 Clinical Study Group. Effects of exenatide (exendin-4) on glycemic control over 30 weeks in sulfonylurea-treated patients with type 2 diabetes. Diabetes Care. 2004 Nov;27(11):2628-35. doi: 10.2337/diacare.27.11.2628. PMID 15504997
- [Derived] Pencek R, Blickensderfer A, Li Y, Brunell SC, Anderson PW. Exenatide twice daily: analysis of effectiveness and safety data stratified by age, sex, race, duration of diabetes, and body mass index. Postgrad Med. 2012 Jul;124(4):21-32. doi: 10.3810/pgm.2012.07.2567. PMID 22913891
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356